CLINICAL TRIAL: NCT00928135
Title: Randomized Controlled Study of Aerosolized Hypertonic Xylitol Versus Hypertonic Saline in Hospitalized Patients With Exacerbation of Cystic Fibrosis
Brief Title: Aerosolized Hypertonic Xylitol Versus Hypertonic Saline in Cystic Fibrosis (CF) Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph Zabner (Other)
Responsible Party: Sponsor-Investigator, Joseph Zabner, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 200901713
Record Dates: First submitted 2009-06-18; First posted 2009-06-25 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Xylitol; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 7% Hypertonic saline (Active Comparator): 5 ml of 7% saline twice daily
  Interventions: Drug: Hypertonic saline
- Hypertonic xylitol (Experimental): 5 ml of 15% xylitol twice daily
  Interventions: Drug: Xylitol

INTERVENTIONS:
Drug: Xylitol — 15% xylitol solution for aerosol; Dosage: 5 ml twice a day (BID)
  Arms: Hypertonic xylitol
Drug: Hypertonic saline — 7% hypertonic saline solution for aerosol; Dosage: 5 ml twice a day (BID)
  Arms: 7% Hypertonic saline

SUMMARY:
Cystic fibrosis (CF) lung disease is characterized by chronic bacterial colonization and recurrent infection of the airways. Lowering the airway surface liquid (ASL) salt concentration has been shown to increase activity of salt sensitive antimicrobial peptides.

Xylitol is a 5-carbon sugar that can lower the ASL salt concentration, thus enhancing innate immunity. In this study, the investigators propose to test the safety and tolerability of aerosolized xylitol used daily for 2 weeks in subjects with cystic fibrosis. In a pilot, 2-week study, 60 subjects with cystic fibrosis with an FEV1(Forced expiratory volume in 1 second ) >30% predicted will be randomized to receive aerosolized 7% hypertonic saline (5 ml) or 15% xylitol, (5 ml) twice a day for 14 days. The primary outcomes will be safety as assessed by FEV1 change from baseline, adverse events and respiratory symptom score. Outcomes for trend in efficacy include density of colonization of sputum, time to next exacerbation, sputum cytokines and revised CF quality of life questionnaire.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) lung disease is characterized by chronic bacterial colonization and recurrent infection of the airways. Disruption of the cystic fibrosis transmembrane conductance regulator chloride channels in subjects with CF results in altered fluid and electrolyte transport across the airway epithelium thereby initiating infections.

These infections eventually destroy the lungs and contribute to significant morbidity and mortality in patients with CF. It is well known that antibacterial activity of innate immune mediators such as lysozyme and beta defensins in human airway surface liquid (ASL) is salt-sensitive; an increase in salt concentration inhibits their activity.

Conversely, their activity is increased by low ionic strength. Lowering the ASL salt concentration and increasing the ASL volume might therefore potentiate innate immunity and therefore decrease or prevent airway infections in subjects with CF.

Xylitol, a five-carbon sugar with low transepithelial permeability, which is poorly metabolized by bacteria can lower the salt concentration of both cystic fibrosis (CF) and non-CF epithelia in vitro. Xylitol is an artificial sweetener that has been successfully used in chewing gums to prevent dental caries; it has been used as an oral sugar substitute without significant adverse effects. It has also been shown to decrease the incidence of acute otitis media by 20-40%; nasal application to normal human subjects was found to decrease colonization with coagulase negative staphylococcus. We found that aerosolized iso-osmolar xylitol was safe in mice, healthy volunteers and stable subjects with CF when administered over a single day. In a recent study, we observed that single doses of 10% followed by 15% xylitol was well tolerated by subjects with cystic fibrosis who were stable. In this pilot study we propose to test the hypothesis that aerosolized hypertonic xylitol given daily for 2 weeks, will be safe and well tolerated and potentially lower the density of colonization in subjects with CF compared to hypertonic saline. We chose hypertonic concentration of xylitol to be comparable in part to hypertonic saline which is being offered as a routine treatment in hospitalized patients with CF exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CF (medical record evidence of CFTR(Cystic fibrosis transmembrane conductance regulator) mutation or sweat chloride test or nasal voltage difference, and 1 or more clinical findings of CF),
* Age 12 or greater
* FEV1 > 30% predicted(within the last 14 days and oxygen saturation > 90% on FiO2(fraction of inspired oxygen) ≤ 50%,
* Admitted for an exacerbation,
* Use of effective contraception in women,
* Able to provide written informed consent.

Exclusion Criteria:

* Pregnancy,
* History of asthma based on methacholine challenge or bronchial hyperresponsiveness on PFTS(Pulmonary Function Test),
* Hemoptysis more than 60 mL within the last 30 days,
* Use of any investigational study drug within the last 30 days,
* Initiation of hypertonic saline within the last 30 days,
* A serum creatinine 2 mg/dl or more
* Active malignancy in the last year
* Antibiotics for CF exacerbation as an outpatient in the last 2 weeks
* B cepacia colonization
* Waiting list for lung transplant
* Lack of FEV1 data from the last 14 days
* Previous participation in this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zabner, M.D., Principal Investigator — PMID: 16781897; Lakshmi Durairaj, M.D., Study Director — PMID: 16781897; Jan L Launspach, R.N., CCRC, Study Chair — PMID: 16781897
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Durairaj L, Launspach J, Watt JL, Mohamad Z, Kline J, Zabner J. Safety assessment of inhaled xylitol in subjects with cystic fibrosis. J Cyst Fibros. 2007 Jan;6(1):31-4. doi: 10.1016/j.jcf.2006.05.002. Epub 2006 Jun 15. PMID 16781897
- [Background] Durairaj L, Neelakantan S, Launspach J, Watt JL, Allaman MM, Kearney WR, Veng-Pedersen P, Zabner J. Bronchoscopic assessment of airway retention time of aerosolized xylitol. Respir Res. 2006 Feb 16;7(1):27. doi: 10.1186/1465-9921-7-27. PMID 16483382
- [Background] Brown CL, Graham SM, Cable BB, Ozer EA, Taft PJ, Zabner J. Xylitol enhances bacterial killing in the rabbit maxillary sinus. Laryngoscope. 2004 Nov;114(11):2021-4. doi: 10.1097/01.mlg.0000147939.90249.47. PMID 15510034
- [Background] Durairaj L, Launspach J, Watt JL, Businga TR, Kline JN, Thorne PS, Zabner J. Safety assessment of inhaled xylitol in mice and healthy volunteers. Respir Res. 2004 Sep 16;5(1):13. doi: 10.1186/1465-9921-5-13. PMID 15377394
- [Background] Zabner J, Seiler MP, Launspach JL, Karp PH, Kearney WR, Look DC, Smith JJ, Welsh MJ. The osmolyte xylitol reduces the salt concentration of airway surface liquid and may enhance bacterial killing. Proc Natl Acad Sci U S A. 2000 Oct 10;97(21):11614-9. doi: 10.1073/pnas.97.21.11614. PMID 11027360
- [Derived] Holliday ZM, Launspach JL, Durairaj L, Singh PK, Zabner J, Stoltz DA. Effects of Tham Nasal Alkalinization on Airway Microbial Communities: A Pilot Study in Non-CF and CF Adults. Ann Otol Rhinol Laryngol. 2022 Sep;131(9):1013-1020. doi: 10.1177/00034894211051814. Epub 2021 Oct 21. PMID 34674574
- [Derived] Hurley MN, Smith S, Forrester DL, Smyth AR. Antibiotic adjuvant therapy for pulmonary infection in cystic fibrosis. Cochrane Database Syst Rev. 2020 Jul 16;7(7):CD008037. doi: 10.1002/14651858.CD008037.pub4. PMID 32671834
- [Derived] Singh S, Hornick D, Fedler J, Launspach JL, Teresi ME, Santacroce TR, Cavanaugh JE, Horan R, Nelson G, Starner TD, Zabner J, Durairaj L. Randomized controlled study of aerosolized hypertonic xylitol versus hypertonic saline in hospitalized patients with pulmonary exacerbation of cystic fibrosis. J Cyst Fibros. 2020 Jan;19(1):108-113. doi: 10.1016/j.jcf.2019.06.016. Epub 2019 Jul 18. PMID 31327670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. subject screen failed due to intolerance to hypertonic saline
  2. subjects failed xylitol trial inhalation
Groups:
- 7% Hypertonic Saline: 5 ml of 7% saline twice daily
  Saline: 7% hypertonic saline solution for aerosol; Dosage: 5 ml twice a day (BID)
Period: Overall Study
Arm/Group | 7% Hypertonic Saline | Hypertonic Xylitol
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypertonic Saline: 7% hypertonic saline given twice daily for 14 days
- Xylitol: Xylitol given twice daily for 14 days
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline | Xylitol | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (12.8) | 29.7 (12.3) | 30.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 17 | 15 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 30 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Forced Expiratory volume % predicted [Mean (Standard Deviation); unit: Percentage predicted] | 53.3 (18.8) | 58.8 (20.1) | 56.1 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 Percentage Predicted From Baseline
Description: Change in lung function (forced expiratory volume in 1 second) between baseline and Day 14
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: percentage of predicted
Arm/Group | 7% Hypertonic Saline | Hypertonic Xylitol
Number analyzed (Participants) | 29 | 30
percentage of predicted | 11.8 [8.1 to 15.5] | 8.8 [4.7 to 12.9]

2. Secondary Outcome: Density of Colonization of Pseudomonas Aeruginosa Per Gram of Sputum
Description: Mean difference from baseline of Sputum density expressed as log colony forming units between baseline and Day 14
Time Frame: 14 days
Population: Subjects who were able to produce sputum at baseline and day 14
Measure: Mean (95% Confidence Interval); unit: log CFU/ml
Arm/Group | 7% Hypertonic Saline | Hypertonic Xylitol
Number analyzed (Participants) | 18 | 22
log CFU/ml | -1.4 [-2.8 to 0.1] | -0.9 [-2.3 to 0.4]

3. Secondary Outcome: Exacerbations During 6 Months Follow-up
Description: numbers of subjects that experienced an exacerbation during the 6 months follow-up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 7% Hypertonic Saline | Hypertonic Xylitol
Number analyzed (Participants) | 29 | 30
Participants | 15 | 11

ADVERSE EVENTS:
Time Frame: For the duration of the study treatment (up tp 14 days) and Up to 7 days after last study drug inhalation for a total of up to 21 days
Arm/Group | 7% Hypertonic Saline | Hypertonic Xylitol
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/29 | 0/30
Other Adverse Events (participants affected / at risk) | 11/29 | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7% Hypertonic Saline (N=29) | Hypertonic Xylitol (N=30)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0) — DIOS is a common problem among CF patients and was deemed unrelated to the study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7% Hypertonic Saline (N=29) | Hypertonic Xylitol (N=30)
abnormal laboratory values (Hepatobiliary disorders) | 5 (5) | 4 (4) — abnormal liver function tests
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — wheezing
Bowel obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Influenza like illness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT00928135/Prot_SAP_000.pdf